CLINICAL TRIAL: NCT05317559
Title: Cardiometabolic Outcomes With Light Exposure During Sleep
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Phyllis Zee, Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: STU00094737
Record Dates: First submitted 2021-12-09; First posted 2022-04-08 (Actual); Last update posted 2022-04-08 (Actual); Status verified 2022-03

CONDITIONS: Light
Keywords: light; sleep; metabolism; sympathetic nervous system; insulin resistance
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- room light (Experimental): The room light condition (n=10) included one night of sleep in dim light (< 3 lux) followed by one night of sleep with overhead room lighting (100 lux).
  Interventions: Behavioral: room light
- dim light (No Intervention): The dim light condition (n=10) included two consecutive nights of sleep in dim light.

INTERVENTIONS:
Behavioral: room light — The room light condition (n=10) included one night of sleep in dim light (< 3 lux) followed by one night of sleep with overhead room lighting (100 lux). The dim light condition (n=10) included two consecutive nights of sleep in dim light.
  Arms: room light

SUMMARY:
This study tested the hypothesis that acute exposure to light during nighttime sleep adversely affects cardiometabolic function.

DETAILED DESCRIPTION:
This study tested the hypothesis that acute exposure to light during sleep adversely affects next morning glucose homeostasis and whether this effect occurs via reduced sleep quality, melatonin suppression, or sympathetic nervous system (SNS) activation during sleep. Twenty young adults participated in this parallel-group study design. The room light condition (n=10) included one night of sleep in dim light (< 3 lux) followed by one night of sleep with overhead room lighting (100 lux). The dim light condition (n=10) included two consecutive nights of sleep in dim light.

ELIGIBILITY:
Inclusion Criteria:

* healthy adults
* ages 18-40 years
* habitual sleep duration of 6.5-8.5 hours
* habitual sleep onset of 9:00 pm-1:00 am

Exclusion Criteria:

* any sleep disorder as assessed by history and screening questionnaires for obstructive sleep apnea (Berlin) and excessive daytime sleepiness (ESS >12), and by PSG to exclude sleep apnea (apnea hypopnea index ≥ 15), periodic leg movements (movement arousal index ≥ 15), or REM sleep behavior disorder;
* history of a cognitive or neurological disorder;
* history of a major psychiatric disorder, including but not limited to mood/anxiety, eating, and alcohol/substance abuse disorders;
* depressed mood (Beck Depression Inventory II score ≥ 20);
* diabetes or other endocrine disorders;
* any gastrointestinal disease requiring dietary adjustment;
* blindness or significant vision loss;
* any unstable or serious medical conditions;
* current or recent (within the past month) of psychoactive, hypnotic, stimulant or analgesic medications;
* shift work or other types of self-imposed irregular sleep schedules;
* obesity (body mass index > 30 kg/m2);
* history of habitual smoking (6 or more cigarettes per week) or drinking (7 or more alcoholic beverages per week) or caffeine consumption greater than 300 mg per day;
* current use of light therapy;
* use of any other legal or illicit substance that may affect sleep and/or appetite;
* allergy to heparin.
* Due to the metabolic stress associated with pregnancy and breastfeeding, patients who were pregnant or breastfeeding were also excluded.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Matsuda Index | Day 2
  OGTT
Matsuda Index | Day 3
  OGTT
HOMA-IR | Day 2
  Fasting
HOMA-IR | Day 3
  Fasting

SECONDARY OUTCOMES:
Sleep Stages | Night 1
  Stage N1, N2, N3
Sleep Stages | Night 2
  Stage N1, N2, N3
Sleep Stages | Night 3
  Stage N1, N2, N3
Heart Rate | Night 2
  beat to beat
Heart Rate | Night 3
  beat to beat
Blood pressure | Day 2
  diastolic/systolic
Blood pressure | Day 3
  diastolic/systolic
Slow Wave Activity | Night 1
  Spectral power in the Slow Wave Activity (0.5 to 4 Hz)
Slow Wave Activity | Night 2
  Spectral power in the Slow Wave Activity (0.5 to 4 Hz)
Slow Wave Activity | Night 3
  Spectral power in the Slow Wave Activity (0.5 to 4 Hz)

OTHER OUTCOMES:
Melatonin | Day 2
  pg/ml
Melatonin | Day 3
  pg/ml
subjective sleepiness | Day 2
  sleepiness level
subjective sleepiness | Day 3
  sleepiness level
hunger | Day 2
  hunger level
hunger | Day 3
  hunger level

IPD SHARING:
Plan to Share IPD: Yes
De-identified data to support the findings of the study are available in Arch, the open access Northwestern University Institutional Repository (https://doi.org/10.21985/n2-9zrx-ev05)